CLINICAL TRIAL: NCT00224328
Title: Measurement of Tissue Oxygen Saturation in Chronic Critical Limb Ischemia: A Phase Iia, Non-Randomized Study Using the ODISsey Tissue Oximeter to Evaluate the Correlation Between Tissue Oxygen Saturation and Symptom Resolution in Patients With Chronic Critical Limb Ischemia Undergoing Treatment Interventions
Brief Title: Measurement of Tissue Oxygen Saturation in Chronic Critical Limb Ischemia
Status: Terminated | Type: Observational
Why Stopped: The results were not able to be consistantly reproduced. Thus the trial was terminated
Sponsor: ViOptix Canada (Industry)
Other Study IDs: VIO-UHN-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Tissue Oxygen Saturation; Peripheral Arterial Disease; Critical Limb Ischemia; Near-infrared Spectroscopy
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: ODISsey Tissue Oximeter

SUMMARY:
Near-infrared spectroscopy can be used to determine the relative oxygen saturation in tissues up to 2cm below the skin. It has been investigated, with success, in cerebral, gastrointestinal, and muscle tissue, and shows promise in numerous indications involving tissue ischemia. In the current study, we propose to examine one hundred patients requiring either bypass or angioplasty due to chronic critical limb ischemia resulting from peripheral arterial disease. We intend to challenge patients before and after the intervention, using either an inflated blood pressure cuff or toe raises, to determine if oxygen saturation recovery time in the affected limb is correlated with symptom resolution (i.e. treatment success). Near-infrared spectroscopy will be performed using the ODISsey tissue oximeter developed by ViOptix, Inc. The proposed study will take approximately one year to complete enrolment, and has a follow-up period of 6 months post-intervention.

Study Hypothesis: Knowledge of tissue oxygen saturation enhances clinical decision making in patients with chronic critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* PAD
* Chronic Critical Limb Ischemia
* requiring surgical intervention
* able to give informed consent

Exclusion Criteria:

* emergent/urgent requirement for surgical intervention
* requiring surgical intervention due to acute traumatic injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-08; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lindsay, FRCSC, FACS, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kooijman HM, Hopman MT, Colier WN, van der Vliet JA, Oeseburg B. Near infrared spectroscopy for noninvasive assessment of claudication. J Surg Res. 1997 Sep;72(1):1-7. doi: 10.1006/jsre.1997.5164. PMID 9344707
- [Background] Simonson SG, Piantadosi CA. Near-infrared spectroscopy. Clinical applications. Crit Care Clin. 1996 Oct;12(4):1019-29. doi: 10.1016/s0749-0704(05)70290-6. PMID 8902382
- [Background] Mancini DM, Bolinger L, Li H, Kendrick K, Chance B, Wilson JR. Validation of near-infrared spectroscopy in humans. J Appl Physiol (1985). 1994 Dec;77(6):2740-7. doi: 10.1152/jappl.1994.77.6.2740. PMID 7896615
- [Background] Mohler LR, Styf JR, Pedowitz RA, Hargens AR, Gershuni DH. Intramuscular deoxygenation during exercise in patients who have chronic anterior compartment syndrome of the leg. J Bone Joint Surg Am. 1997 Jun;79(6):844-9. doi: 10.2106/00004623-199706000-00007. PMID 9199381
- [Background] Cheatle TR, Potter LA, Cope M, Delpy DT, Coleridge Smith PD, Scurr JH. Near-infrared spectroscopy in peripheral vascular disease. Br J Surg. 1991 Apr;78(4):405-8. doi: 10.1002/bjs.1800780408. PMID 2032098
- [Background] Jarm T, Kragelj R, Liebert A, Lukasiewitz P, Erjavec T, Preseren-Strukelj M, Maniewski R, Poredos P, Miklavcic D. Postocclusive reactive hyperemia in healthy volunteers and patients with peripheral vascular disease measured by three noninvasive methods. Adv Exp Med Biol. 2003;530:661-9. doi: 10.1007/978-1-4615-0075-9_66. PMID 14562764
- [Background] Lee BY, Ostrander E, Karmakar M, Frenkel L, Herz B. Noninvasive quantification of muscle oxygen in subjects with and without claudication. J Rehabil Res Dev. 1997 Jan;34(1):44-51. PMID 9021624
- [Background] 8. TransAtlantic Inter-Society Consensus Document. (living document, 1999) Management of Peripheral Arterial Disease: Critical Limb Ischemia. http://www.tasc-pad.org/ Arterial Disease. J Vasc Surg; Oct; 38(4): 724-9.
- [Background] Reifsnyder T, Grossman JP, Leers SA. Limb loss after lower extremity bypass. Am J Surg. 1997 Aug;174(2):149-51. doi: 10.1016/s0002-9610(97)90074-x. PMID 9293832
- [Background] Troeng T, Bergqvist D, Janson L. Incidence and causes of adverse outcomes of operation for chronic ischaemia of the leg. Eur J Surg. 1994 Jan;160(1):17-25. PMID 8186308